CLINICAL TRIAL: NCT06190717
Title: Maturation of Arteriovenous Fistula With Automated Sonography Assessments Trial
Acronym: MAFASA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonavex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAFASA-2023
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Diabetes; End Stage Renal Disease
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Diagnostic Arm (Experimental): All subjects will have the EchoMark implanted. Subjects will be assessed every 2 weeks (+/- 1 week) (but no more frequently than weekly) with the EchoSure system until fistula maturation occurs and/or permanent access use is achieved.
  Interventions: Device: EchoMark/EchoSure
- Standard of Care (Active Comparator): Subjects will be evaluated per KDOQI guidelines (with physical examination at approximately 2 weeks (+/- 1 week) and between 4 and 6 weeks (+/- 1 week)). If evaluation yields abnormal findings, subjects will receive a Duplex ultrasound assessment (DUS). All SOC Arm subjects will be followed per the institution's standard of care until fistula maturation occurs and/or permanent access use is achieved but no more frequently than once per month.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Device: EchoMark/EchoSure — Subjects assigned to the Diagnostic Arm will have the EchoMark implanted at the time of AVF creation. The subject will return every 2 weeks for a follow-up assessment to include an EchoSure scan until fistula maturation and/or permanent access use is achieved. The EchoSure scans are to be reviewed by the investigator(s) or delegated study staff and aid in the determination when a further assessment, including a physical exam, is required to determine cannulation clearance or if an intervention(s) may be required to prevent failure of fistula maturation. All physical exams will include assessing the fistula for bruit and thrill. The subject's medical history will be reviewed at each visit and will include all interventions, cannulation attempts, and adverse event reporting.
  Arms: Diagnostic Arm
Procedure: Standard of Care — Subjects are assessed using standard of care per KDOQI guidelines, which includes a physical exam at the 2-week follow-up visit and at the 4-6-week follow-up visit. All follow-up visits will include an assessment of adverse events and medical history review to include all interventions, cannulation attempts, and laboratory results. If evaluation yields an abnormal finding, subjects will undergo a Duplex ultrasound assessment and treatment under the institution's standard of care. All SOC Arm subjects will be followed per the institution's standard of care until fistula maturation occurs and/or permanent access use is achieved but no more frequently than once per month.
  Arms: Standard of Care

SUMMARY:
This is a prospective, multi-center, two-arm, randomized trial to quantify the performance of the EchoMark®/EchoSure® System for AVF diagnostic ultrasound when used under a protocol of biweekly use for assessing fistula maturation and reducing time to Clinical Maturation.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females ≥ 18 years of age but < 85 years of age at the time of informed consent.
* Subject is able and willing to provide written informed consent prior to receiving any non-standard of care, protocol specific procedures.
* Subject is willing and capable of complying with all required follow-up visits.
* Subject and/or Care Team agree that the distance and transportation resources from the patient's home to the clinic are reasonable for study participation and compliance.
* Subject has an estimated life expectancy > 18 months.
* Subject is ambulatory (cane or walker are acceptable).
* CKD Stage 5 (eGFR less than 10) or ESRD subjects presenting for upper arm autologous arteriovenous fistula creation that is not transposed for hemodialysis access.
* Subjects who are currently on dialysis through a CVC or who imminently require dialysis (GFR <10).
* Vein diameter ≥ 2.5 mm at the antecubital fossa per vein mapping.
* Artery diameter ≥ 2.5 mm per vein mapping.
* Subject is not participating in another investigational clinical trial that has not met its primary end point. Participation in post-market registry is acceptable.

Exclusion Criteria:

* CKD Stage 1-4 or subjects that do not require upper arm autologous arteriovenous fistula creation for hemodialysis access.
* Subject has history of Steal Syndrome.
* Subject who is immunocompromised or immunosuppressed.
* Subject has had three previous failed AV fistulae for hemodialysis access.
* Subjects expecting to undergo major surgery within 60 days from the EchoMark implantation.
* Known or suspected active infection on the day of the index procedure.
* Subjects who had infection(s) in the 30-day window prior to EchoMark placement to reduce the likelihood of partially treated infections that can seed the device and fistula.
* Subjects with diagnosed bleeding disorder, thrombocytopenia (platelet count <50,000), hypercoagulability, and history of recurrent deep vein thrombosis not related to AV access.
* Subjects with active malignancy.
* Subjects with a history of poor compliance with the dialysis protocol.
* Subjects with a known or suspected allergy to any of the device materials.
* Subjects with an existing fistula or graft.
* Subjects who are anticipated to convert to peritoneal dialysis or undergo a transplant within 6 months.
* Subjects who are pregnant, planning on becoming pregnant, or are breast feeding.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 6 months
  Freedom from the following through 6 months as adjudicated by the CEC:
  1. Clinically significant misplacement or migration of the EchoMark implant.
  2. Vessel or tissue injury caused by the EchoMark implant procedure of the implant over time, requiring surgical intervention.
  3. Infection of tissues surrounding the EchoMark implant requiring IV/
  4. Complication requiring explantation of the EchoMark implant.
Primary Effectiveness Endpoint | 6 months
  Time to clinical maturation

SECONDARY OUTCOMES:
Difference between EchoSure and Duplex Flow Measurements | 6 Months
  Difference between log10-transformed EchoSure and Duplex flow measurements of blood flow for assessment of measurement agreement in the diagnostic arm.
EchoSure Depth Comparison | 6 Months
  Difference between EchoSure and CoreLab measurements of depth for assessment of measurement agreement in the diagnostic arm.
EchoSure Diameter Comparison | 6 Months
  Difference between EchoSure and CoreLab measurement of diameter for assessment of measurement agreement in the diagnostic arm.
EchoMark/EchoSure System Technical Success | 4 Months
  Technical Success defined as the successful implantation of the EchoMark implant and the ability to complete each scan to determine the blood flow, diameter, and depth measurements at the EchoMark using the EchoSure diagnostic ultrasound system from baseline to Clinical Maturation, fistula failure, or 4 months, whichever is sooner.
CVC Removal | 6 Months
  Time to CVC removal by subject group
Rate of Hospitalization | 6 Months
  Rate of hospitalization(s) by subject group from baseline to Clinical Maturation.
AV Fistula Maturation Rate | 6 Months
  Percent of AVFs created that mature by 180 days by subject group.
Total Cost of Care | 6 Months
  Total cost of care, defined by National average Medicare payment rate (facility and professional fees) for procedures and care provided to subject by subject group from baseline to Clinical Maturation.
Freedom from Events through 30 and 90 Days | 30 Days and 90 Days
  Freedom from the following through 30 and 90 days from the baseline procedure as adjudicated by the CEC:
  1. Clinically significant misplacement or migration of the EchoMark implant.
  2. Vessel or tissue injury caused by the EchoMark implant procedure of the implant over time, requiring surgical intervention.
  3. Infection of tissues surrounding the EchoMark implant requiring IV antibiotic treatment.
  4. Complication requiring explantation of the EchoMark implant.

OTHER OUTCOMES:
Hierarchical Composite 1 | 6 Months
  Hierarchical composite of the DIAG arm and SOC arm comparing occurrences of:
  Fistula creation success.
Hierarchical Composite 2 | 6 Months
  Hierarchical composite of the DIAG arm and SOC arm comparing occurrences of:
  Alive through 180 days.
Hierarchical Composite 3 | 6 Months
  Hierarchical composite of the DIAG arm and SOC arm comparing occurrences of:
  Freedom from SAE with 180 days (severity as a tie-breaker for SAEs with matching adverse event term)
Hierarchical Composite 4 | 6 Months
  Hierarchical composite of the DIAG arm and SOC arm comparing occurrences of:
  Earlier time to AV fistula Clinical Maturation with 180 days.
Comparison of Composite and Stratified MAE Rates | 6 Months and 12 Months
  Comparison of composite and stratified MAE rates for both subject groups at 6 months and end of study. MAEs are adjudicated by the CEC and defined as any of the following:
  1. Clinically significant misplacement or migration of the EchoMark implant.
  2. Vessel or tissue injury caused by the EchoMark implant procedure or the implant over time, requiring surgical intervention.
  3. Complication requiring explantation of the EchoMark implant.
  4. Clinically significant surgical complications (seroma, edema, hematoma, bleeding), excluding expected resorption response visible as hypoechoic region on B-mode ultrasound.
  5. Infection requiring IV antibiotic treatment. Pseudoaneurysm.
  6. Thrombosis of the AVF circuit that requires an intervention (surgical or endovascular).
  7. Steal Syndrome.
Comparision of Implant and Procedure Related Adverse Events | 6 Months and 12 Months
  Comparison of all stratified implant and procedure related AE (as adjudicated by the CEC) rates between subject groups at 6 months and end of study.
Clinical Maturation | 3 Months, 4 Months, 5 Months, and 6 Months
  Percent of subjects that have reached Clinical Maturation (as adjudicated by the CEC) for each subject group at 90 days, 120 day, 150 days, and 180 days.
Cannulation Complication Rates | 12 Months
  Comparison of composite and stratified cannulation complication (as adjudicated by the CEC) rates between subject groups for the following AEs:
  1. Infection due to cannulation.
  2. Thrombosis due to hematoma.
  3. Any other AE determined by the CEC to be cannulation related.
Time to Clinical Maturation for Procedure and Device Related Events | 6 Months
  Distribution of time to Clinical Maturation for both groups for each of the following procedure and device related categories presented as violin/box plots:
  1. Clinically significant misplacement or migration of the EchoMark implant.
  2. Vessel or tissue injury caused by the EchoMark implant procedure or the implant over time, requiring surgical intervention.
  3. Clinically significant surgical complications (seroma, edema, hematoma, bleeding), excluding expected resorption response visible as hypoechoic region on B-mode ultrasound.
  4. Infection requiring IV antibiotic treatment.
  5. Pseudoaneurysm.
  6. Thrombosis of AVF circuit requiring an intervention (surgical or endovascular).
  7. Steal Syndrome.
  8. No SAE.
Primary Functional Patency | 6 Months
  Primary functional patency at 6 months (as adjudicated by the CEC) defined as freedom from intervention on the AVF after maturation.
Secondary Function Patency | 6 Months
  Secondary functional patency at 6 months (as adjudicated by the CEC) is defined as freedom from abandonment of the AVF after maturation.
Time to Clinical Maturation | 6 Months
  Time to Clinical Maturation (as adjudicated by the CEC) defined as the time from initial fistula creation to Clinical Maturation.
Time to Clinical Maturation for Each Fistula | 6 Months
  Time to Clinical Maturation (as adjudicated by the CEC) for each new fistula defined as the time from new fistula creation to Clinical Maturation.
Technical Success Cannulation Scans | 4 Months
  Rate of cannulation zone technical success rate defined as the ability to complete each scan to determine the diameter, and depth measurements at the proximal, mid, and distal segments of the fistula using the EchoSure diagnostic ultrasound system from the 2-week follow-up to Clinical Maturation, or 4 months, whichever is sooner.
EchoSure Diameter and Depth Comparison in Cannulation Zone | 6 Months
  Agreement of EchoSure diameter and depth results from the cannulation zone at the 6-week follow-up compared to the CoreLab measured diameter and depth results in the DIAG arm.
Intervention to Assist Maturation Rate | 6 Months
  Surgical or Endovascular Interventions to Assist Maturation defined as the difference between groups in the proportion of subjects with surgical or endovascular interventions to assist maturation.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Trinity Research Group, Dothan, Alabama
  - Southwest Kidney Institute, Phoenix, Arizona
  - AKDHC Medical Research Services, Phoenix, Arizona
  - AKDHC Center Tucson, Tucson, Arizona
  - Orlando Health Heart and Vascular Institute, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Kansas Nephrology Research Institute, Wichita, Kansas
  - Boston Medical Center, Boston, Massachusetts
  - MSU Health Care Heart and Vascular, Lansing, Michigan
  - Capital Medical Center, Pennington, New Jersey
  - Northwell Health, New Hyde Park, New York
  - Atrium Health, Concord, North Carolina
  - Prisma Health, Greenville, South Carolina
  - Medical University of South Carolina Health Orangeburg, Orangeburg, South Carolina
  - Galen Medical Group, Chattanooga, Tennessee
  - Fresenius Vascular Care Memphis MSO, Memphis, Tennessee
  - Baylor Scott & White Heart and Vascular Hospital, Dallas, Texas
  - Aqua Research Institute Llc, Houston, Texas
  - Physicians Care of Virginia, Roanoke, Virginia
  - Sentara Health, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No